CLINICAL TRIAL: NCT06380036
Title: a Comparison of the Recurrence of Fistula in Ano After Video Assisted Fistulectomy VS. Loose Seton in Surgical Patients Having Fistula in Ano
Brief Title: Two Approaches to Lower the Chances of Recurrence of Anal Fistula After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sairah Sadaf (Other Government)
Responsible Party: Sponsor-Investigator, Sairah Sadaf, Classified Consultant, Sheikh Zayed Medical College
Organization: Sheikh Zayed Medical College (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003AEstb/EC/01/2022
Record Dates: First submitted 2024-04-15; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Fistula in Ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- seton (Experimental): loose seton will be placed in the pts with fistula in ano. All patients in Group A underwent the loose seton technique. The procedures were performed in the operating room with the patient in the lithotomy position. Probing of the fistula tract was done with a metallic malleable probe. The incision was given from the external opening of the fistula to the anal verge, involving the skin, subcutaneous tissue, superficial part of the external sphincter, and superficial part of the internal sphincter. After the insertion of loose Seton, a non-absorbable suture was left loosely and kept in situ for three months.
  Interventions: Procedure: video assisted fistula tract surgery
- VAAFTS (Experimental): In group B, video-assisted fistula tract surgery (VAAFTS) was performed. The patients were positioned in the lithotomy position. The fistuloscope was then introduced into the external opening and the procedure was performed, except for the closure of the internal opening, which was performed with either a "figure of eight" suture or an advancement flap, rather than using a stapler. The tracts were destroyed using electrocautery, the necrotic tissues were removed, and the external openings were cored out and left open for drainage
  Interventions: Procedure: video assisted fistula tract surgery

INTERVENTIONS:
Procedure: video assisted fistula tract surgery — in one group pt recieved VAAFTS
  Other Names: Loose setone

SUMMARY:
A total of 80 patients with complex fistula in ano of both genders were included. All patients in Group A underwent a loose seton technique. In group B, video-assisted fistula tract surgery (VAAFTS) was performed.Twice daily Sitz baths, analgesics, and stool bulking agents (bran) were used in follow-up care. Repeated examinations were carried out every four weeks and recurrence was noted at the end of three months

DETAILED DESCRIPTION:
Patients were equally allocated into two groups i.e. Group A & Group B by lottery method. In both groups, the lower bowel was emptied by an enema about an hour before the operation. All patients in Group A underwent the loose seton technique. The procedures were performed in the operating room with the patient in the lithotomy position. Probing of the fistula tract was done with a metallic malleable probe. The incision was given from the external opening of the fistula to the anal verge, involving the skin, subcutaneous tissue, superficial part of the external sphincter, and superficial part of the internal sphincter. After the insertion of loose Seton, a non-absorbable suture was left loosely and kept in situ for three months.

In group B, video-assisted fistula tract surgery (VAAFTS) was performed. The patients were positioned in the lithotomy position. The fistuloscope was then introduced into the external opening and the procedure was performed, except for the closure of the internal opening, which was performed with either a "figure of eight" suture or an advancement flap, rather than using a stapler. The tracts were destroyed using electrocautery, the necrotic tissues were removed, and the external openings were cored out and left open for drainage. The patients were discharged the day following the procedure. Twice daily Sitz baths, analgesics, and stool bulking agents (bran) were used in follow-up care. Repeated examinations were carried out every four weeks and recurrence was noted at the end of three months. The information (age, gender, duration of disease, BMI, diabetes mellitus, hypertension, place of living, and recurrence) was collected through pre-designed Performa (Annexure I).

ELIGIBILITY:
1. Inclusion Criteria:

   * complex fistula in ano (as per operational definition)
   * with a duration of disease >1 month,
   * either gender
   * history of previous surgery for fistula in ano
2. Exclusion Criteria:

   * Pregnant females
   * bleeding disorder
   * history of pulmonary or systemic tuberculosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
recurrence | one year
  to see whether recurrence occur or not

CONTACTS AND LOCATIONS:
Overall Officials: sairah sadaf, fcps, Principal Investigator — sheikh zayed medical college rhaim yar khan
Locations (1):
- Sheikh Zayed Medical College, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No